CLINICAL TRIAL: NCT01504841
Title: A Phase I/II, Open-Label Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Etravirine (ETR) in Antiretroviral (ARV) Treatment-Experienced HIV-1 Infected Infants and Children, Aged ≥ 2 Months to < 6 Years
Brief Title: Evaluating the Safety and Tolerability of Etravirine in HIV-1 Infected Infants and Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1090; 10850 (Other: DAIDS-ES)
Record Dates: First submitted 2011-12-30; First posted 2012-01-05 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort I: Treatment experienced, 2 to 6 years of age (Experimental): Children in this arm were at least 2 but younger than 6 years of age; they received the study drug etravirine (ETR) together with an optimized background regimen (OBR) consisting of one active boosted protease inhibitor (PI) and at least one other active antiretroviral (ARV) drug.
  Interventions: Drug: Etravirine (ETR)
- Cohort II: Treatment experienced, 1 to 2 years of age (Experimental): Children in this arm were at least 1 but younger than 2 years of age; they received ETR together with an OBR consisting of one active boosted PI and at least one other active ARV drug.
  Interventions: Drug: Etravirine (ETR)
- Cohort III: Treatment experienced, 2 months to 1 year of age (Experimental): Children in this arm were at least 2 months but younger than 1 year of age; they received ETR together with an OBR consisting of one active boosted PI and at least one other active ARV drug.
  Interventions: Drug: Etravirine (ETR)

INTERVENTIONS:
Drug: Etravirine (ETR) — ETR was administered as 25-mg scored tablets and/or 100-mg tablets swallowed whole or dispersed in an appropriate liquid vehicle following a meal. Children took the specified dose orally twice daily within 30 minutes following a meal. Dose was decided according to dosing tables in protocol.

SUMMARY:
Non-nucleoside reverse transcriptase inhibitors (NNRTIs) are widely used as part of combination antiretroviral therapy (ART) for infants and children, but NNRTI resistance is increasing, leading to treatment failure. This study tested the safety, tolerability, and dosing levels of etravirine (ETR), a new NNRTI.

DETAILED DESCRIPTION:
Use of NNRTI-based regimens as initial therapy for HIV-infected children is increasing, especially in areas where newborns exposed to HIV-1 receive single-dose nevirapine (NVP) as part of prevention of mother-to-child transmission (PMTCT) regimens and/or daily NVP for prevention of transmission through breastfeeding. First-generation NNRTIs have a low genetic barrier to the development of resistance; in two of the most widely used NNRTIs, NVP and efavirenz (EFV), even a single amino acid mutation in the virus can lead to a reduction in the drug's effectiveness. Even short-term use of these NNRTIs, including only a single dose of NVP, can cause NNRTI resistance. Second-generation NNRTIs are needed as part of ARV regimens for newly diagnosed infants and children who have been exposed to single-dose NVP or who have failed their current antiretroviral (ARV) regimens. In this study, the second-generation NNRTI ETR was tested for safety, tolerability, and appropriate dosing.

Children were assigned to one of three cohorts based on age:

* Cohort I: At least 2 but younger than 6 years of age
* Cohort II: At least 1 but younger than 2 years of age
* Cohort III: At least 2 months but younger than 1 year of age

Children in all three cohorts were treatment experienced, defined as being on a failing combination ARV regimen (containing at least 3 ARVs) for at least 8 weeks or having a treatment interruption of at least 4 weeks with a history of virologic failure while on a combination ARV regimen (containing at least 3 ARVs).

Children received ETR together with an optimized background regimen (OBR) consisting of at least 2 active agents (a boosted protease inhibitor [PI] and at least 1 additional active ARV drug). OBR were based on clinical status, treatment history, resistance data, and availability of appropriate pediatric dosing and formulations. The children received an oral dose of ETR twice daily.

Most children had 11 visits: at screening, entry (Day 0), Day 14 (intensive pharmacokinetic [PK] visit), and at Weeks 4, 8, 12, 16, 24, 32, 40, and 48. Most visits included a physical exam, giving a medical history, discussion of adherence, and blood and urine collection. The screening and intensive PK visits also included an electrocardiogram (ECG). During the intensive PK visit, the child had blood drawn approximately 7 times over 12 hours. After the Week 48 visit, children entered the long-term follow-up phase of the study and have a visit every 12 weeks for up to 5 years. These follow-up visits included giving a medical history and undergoing a physical exam and blood draw.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection as described in the protocol
* NOTE: Children who were born at or sooner than 37 weeks gestational age must be at least 12 weeks of age and at least 46 weeks post-conceptual age at study entry.
* HIV-1 RNA viral load greater than 1,000 copies/mL (within the previous 90 days prior to screening) and an HIV-1 RNA viral load greater than 1,000 copies/mL at screening
* Treatment-experienced children on a failing combination antiretroviral (ARV) regimen (containing at least three ARVs) for at least 8 weeks; OR, treatment-experienced children on a treatment interruption of at least 4 weeks with a history of virologic failure while on a combination ARV regimen (containing at least three ARVs)
* Ability to swallow etravirine (ETR) whole or dispersed in an appropriate liquid
* Parent or legal guardian able and willing to provide signed informed consent and to have the child followed at the clinic site
* Availability of sufficient active ARV drugs to create an optimized background regimen (OBR) consistent with protocol requirements

Exclusion Criteria:

* Evidence of phenotypic resistance to ETR at screening (phenotypic cutoffs of greater than 10 for loss of sensitivity for cohorts I, II, III)
* Known history of HIV-2 infection in child or child's mother
* Diagnosis of a new Centers for Disease Control (CDC) Stage C (per 1994 Revised Classification System for Human Immunodeficiency Virus Infection in Children Less than 13 Years of Age) criteria or opportunistic or bacterial infection diagnosed within 30 days prior to screening and not considered clinically stable
* Prior history of malignancy
* Any clinically significant diseases (other than HIV infection) or clinically significant findings during the screening medical history or physical examination that in the investigator's opinion would place the child at an unacceptable risk of injury, render the child unable to meet the requirements of the protocol, compromise the outcome of this study, or lead to the child being ineligible for participation
* Current Grade 3 or higher of any of the following laboratory toxicities at screening: neutrophil count, hemoglobin, platelets, aspartate aminotransferase (AST), alanine aminotransferase (ALT), lipase, or serum creatinine.
* Current or anticipated use of any disallowed medications (listed in the protocol)
* Child's family is unlikely to adhere to the study procedures or keep appointments or is planning to relocate to a non-IMPAACT study site during the study
* History of nonadherence with ARV medications that in the investigator's opinion could affect the ability of the child to comply with the protocol/procedures
* Child is currently participating, or has participated within the previous 30 days prior to screening, in a study with a compound or device that is not commercially available
* Grade 3 or higher QTc or PR interval prolongation from the electrocardiogram (ECG) at screening. More information on this criterion can be found in the protocol.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rutstein, MD, Study Chair — Children's Hospital of Philadelphia
Locations (11):
- United States (4):
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
- Brazil (5):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira - UFRJ NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- South Africa (2):
  - Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng
  - Umlazi CRS, Durban, KwaZulu-Natal

REFERENCES:
- [Background] Jittamala P, Puthanakit T, Chaiinseeard S, Sirisanthana V. Predictors of virologic failure and genotypic resistance mutation patterns in thai children receiving non-nucleoside reverse transcriptase inhibitor-based antiretroviral therapy. Pediatr Infect Dis J. 2009 Sep;28(9):826-30. doi: 10.1097/INF.0b013e3181a458f9. PMID 19654564
- [Background] Palumbo P, Lindsey JC, Hughes MD, Cotton MF, Bobat R, Meyers T, Bwakura-Dangarembizi M, Chi BH, Musoke P, Kamthunzi P, Schimana W, Purdue L, Eshleman SH, Abrams EJ, Millar L, Petzold E, Mofenson LM, Jean-Philippe P, Violari A. Antiretroviral treatment for children with peripartum nevirapine exposure. N Engl J Med. 2010 Oct 14;363(16):1510-20. doi: 10.1056/NEJMoa1000931. PMID 20942667
- See also: Description DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004; Clarification, August 2009 — https://rsc.niaid.nih.gov/sites/default/files/table-for-grading-severity-of-adult-pediatric-adverse-events.pdf
- See also: Description Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/sites/default/files/manual-exped-aes-v2_0.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled March 2013, and the final participant was enrolled June 2017. Participants were accrued from a total of 11 sites across Brazil, South Africa, and the USA.
Pre-assignment Details: Participants were stratified into the 3 Cohorts by age group and not randomized. There were no eligibility violations or errors to cohort assignments.
Period: Overall Study
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Started | 20 | 6 | 0 (No enrollments occurred into Cohort 3 during the study.)
Completed | 19 | 5 | 0
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population is defined as having been treated exclusively on the dose determined to be optimal for a given cohort and having either completed 48 weeks of exposure to the study drug or having been classified as a safety failure, due to a study drug related adverse event occurring during the first 48 weeks of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age | Total
Number analyzed (Participants) | 11 | 4 | 0 | 15
Age, Continuous [Median (Full Range); unit: years] | 4 [3 to 5] | 1 [1 to 1] |  | 3.5 [1 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 |  | 7
  Male | 5 | 3 |  | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 |  | 5
  Not Hispanic or Latino | 3 | 1 |  | 4
  Unknown or Not Reported | 4 | 2 |  | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 8 | 4 |  | 12
  White | 1 | 0 |  | 1
  More than one race | 1 | 0 |  | 1
  Unknown or Not Reported | 1 | 0 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 |  | 3
  Brazil | 3 | 1 |  | 4
  South Africa | 6 | 2 |  | 8
Plasma HIV RNA [Count of Participants; unit: Participants]
  <400 copies/ml | 0 | 0 |  | 0
  400 - <5,000 copies/ml | 4 | 1 |  | 5
  5,000 - <10,000 copies/ml | 0 | 0 |  | 0
  10,000 - < 25,000 copies/ml | 2 | 1 |  | 3
  25,000 - < 50,000 copies/ml | 1 | 1 |  | 2
  >=50,000 copies/ml | 4 | 1 |  | 5
CD4 Count [Count of Participants; unit: Participants]
  50 - <200 cells/mm^3 | 1 | 0 |  | 1
  200 - <350 cells/mm^3 | 1 | 0 |  | 1
  350 - <500 cells/mm^3 | 1 | 1 |  | 2
  >=500 cells/mm^3 | 8 | 3 |  | 11
CD4 Percent [Count of Participants; unit: Participants]
  <= 14 % | 1 | 1 |  | 2
  >14 - <25 % | 5 | 1 |  | 6
  >= 25 % | 5 | 2 |  | 7

OUTCOME MEASURES:

1. Primary Outcome: Termination From Treatment Due to a Suspected Adverse Drug Reaction (SADR)
Description: Number (%) of participants who discontinued treatment due to a suspected adverse drug reaction (SADR) by Cohort.
Time Frame: From baseline to occurrence of event, up to Week 48.
Population: Analysis population is defined as having been treated exclusively on the final dose determined to be optimal for a given cohort without adjustments and having either completed 48 weeks of exposure to the study drug or been classified as a safety failure, due to a study drug related adverse event occurring during the first 48 weeks of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Discontinued treatment due to a SADR | 1 | 0 |
  Did not discontinue treatment due to a SADR | 10 | 4 |

2. Primary Outcome: Adverse Events (AEs) of Grade 3 or Higher Severity
Description: Number (%) of participants who experienced a Grade 3 or higher severity adverse event through Week 48 by Cohort, with Clopper-Pearson confidence intervals.
Time Frame: From baseline to occurrence of event, up to Week 48.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Experienced a grade 3+ AE | 4 | 4 |
  Did not experience a grade 3+ AE | 7 | 0 |
Statistical Analysis 1: Comparison: Cohort I: Treatment Experienced, 2 to 6 Years of Age; Test type: Other; % = 36.4, 95% CI 2-sided [10.9 to 69.2] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort I, percentage of participants who experienced a grade 3+ AE
Statistical Analysis 2: Comparison: Cohort II: Treatment Experienced, 1 to 2 Years of Age; Test type: Other; % = 100, 95% CI 2-sided [39.8 to 100] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort II, percentage of participants who experienced a grade 3+ AE

3. Primary Outcome: Death
Description: Number (%) of deaths on study by Cohort.
Time Frame: From baseline to occurrence of event, up to Week 48.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Deaths | 0 | 0 |
  Live participants | 11 | 4 |

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve Over 12 Hours of ETR
Description: Geometric Mean (Standard Deviation) of the area under the plasma concentration-time curve over 12 hours (AUC12h) of ETR.
Time Frame: Pre-dose, 1, 2, 4, 6, 9, and 12 hours post-dose measured at intensive PK visit (within 7-10 days after last dose of study drug administration)
Population: Analysis population is defined as having been treated exclusively on the final dose determined to be optimal for a given cohort without adjustments and having either completed 48 weeks of exposure to the study drug or been classified as a safety failure. They must also be considered PK evaluable by the study team; 1 Participant in Cohort 1 is not.
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age
Number analyzed (Participants) | 10 | 4
ng*h/mL | 5512.85 (3615.36) | 4821.76 (3167.11)

5. Secondary Outcome: AEs of Grade 3 or Higher Severity Judged to be at Least Possibly Attributable to the Study Medications
Description: Number (%) of Participants with AEs of Grade 3 or higher severity judged, by the Study Team, to be at least possibly attributable to the study medications by Cohort, including Clopper-Pearson confidence intervals.
Time Frame: From baseline to occurrence of event, up to Week 48.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Had a grade 3+ AE related to study drug | 2 | 0 |
  Had no grade 3+ AE related to study drug | 9 | 4 |
Statistical Analysis 1: Comparison: Cohort I: Treatment Experienced, 2 to 6 Years of Age; Test type: Other; % = 18.2, 95% CI 2-sided [2.5 to 51.8] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort I, percentage of participants who experienced a grade 3+ AE at least possibly related to study medications
Statistical Analysis 2: Comparison: Cohort II: Treatment Experienced, 1 to 2 Years of Age; Test type: Other; % = 0, 95% CI 2-sided [0 to 60.2] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort II, percentage of participants who experienced a grade 3+ AE at least possibly related to study medication

6. Secondary Outcome: HIV-1 RNA Virologic Failure Status at Weeks 24 and 48
Description: Number (%) of participants with confirmed Virologic Failure, defined as: failure to suppress plasma HIV-1 RNA to fewer than 400 copies/ml and failure to achieve at least a 2-log10 reduction (from baseline) in HIV-1 RNA at Weeks 24 or 48, by Cohort, with Clopper-Pearson confidence intervals. The initial HIV-1 RNA results that met the Virologic Failure definition were each confirmed by a second result obtained within 1 to 4 weeks of the initial result obtained at Week 24 and/or 48.
Time Frame: Baseline, Week 24, and Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Week 24: Virologic Failure | 2 | 1 |
  Week 24: No Virologic Failure | 9 | 3 |
  Week 48: Virologic Failure | 3 | 3 |
  Week 48: No Virologic Failure | 8 | 1 |
Statistical Analysis 1: Comparison: Cohort I: Treatment Experienced, 2 to 6 Years of Age; Week 24 time point; Test type: Other; % = 18.2, 95% CI 2-sided [2.3 to 51.8] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort I Week 24, percentage of participants who experienced Virologic Failure
Statistical Analysis 2: Comparison: Cohort II: Treatment Experienced, 1 to 2 Years of Age; Week 24 time point; Test type: Other; % = 25, 95% CI 2-sided [0.6 to 80.6] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort II Week 24, percentage of participants who experienced Virologic Failure
Statistical Analysis 3: Comparison: Cohort I: Treatment Experienced, 2 to 6 Years of Age; Week 48 time point; Test type: Other; % = 27.3, 95% CI 2-sided [6 to 61] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort I Week 48, percentage of participants who experienced Virologic Failure
Statistical Analysis 4: Comparison: Cohort II: Treatment Experienced, 1 to 2 Years of Age; Week 48 time point; Test type: Other; % = 75, 95% CI 2-sided [19.4 to 99.4] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort II Week 48, percentage of participants who experienced Virologic Failure

7. Secondary Outcome: Treatment Discontinued Due to Toxicity or Virologic Failure
Description: Number (%) of participants who discontinued study treatment (ETR) due to a toxicity or Virologic Failure (VF), by Cohort.
Time Frame: From baseline to occurrence of event, up to Week 48.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Discontinued Treatment due to VF | 1 | 0 |
  Did not discontinue treatment due to VF | 10 | 4 |

8. Secondary Outcome: Change in Optimized Background Regimen Due to Virologic Failure
Description: Number (%) of participants who initiated a change in their optimized background regimen (OBR) due to virologic failure, by Cohort.
Time Frame: Measured at entry and at Weeks 8, 12, 24, and 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Changed OBR due to Virologic Failure | 0 | 0 |
  Did not change OBR due to Virologic Failure | 11 | 4 |

9. Secondary Outcome: New Onset Opportunistic Infection (OI) or AIDS Diagnosis
Description: Number (%) of participants with a new onset opportunistic infection (OI) or AIDS diagnosis, by Cohort.
Time Frame: From baseline to occurrence of event, up to Week 48.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Had a new OI | 0 | 0 |
  Had no new OIs | 11 | 4 |

10. Secondary Outcome: Decline in Absolute CD4 Percent of Greater Than 5 Percent Any Time After 12 Weeks of Therapy
Description: Number (%) of participants with a >5% decline in absolute CD4 percent from baseline at weeks 12, 24, and 48, by Cohort, including Clopper-Pearson confidence intervals.
Time Frame: Measured at baseline and at Weeks 12, 24, and 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age | Cohort III: Treatment Experienced, 2 Months to 1 Year of Age
Number analyzed (Participants) | 11 | 4 | 0
Participants
  Week 12: >5% decline in CD4 % from baseline | 1 | 2 |
  Week 12: Increase or <5% decline in CD4 % from baseline | 10 | 2 |
  Week 24: >5% decline in CD4 % from baseline | 1 | 1 |
  Week 24: Increase or <5% decline in CD4 % from baseline | 10 | 3 |
  Week 48: >5% decline in CD4 % from baseline | 2 | 2 |
  Week 48: Increase or <5% decline in CD4 % from baseline | 9 | 2 |
Statistical Analysis 1: Comparison: Cohort I: Treatment Experienced, 2 to 6 Years of Age; Week 12 time point; Test type: Other; % = 9.1, 95% CI 2-sided [0.2 to 41.3] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort I Week 12, percentage of participants with a >5% decline in absolute CD4 %
Statistical Analysis 2: Comparison: Cohort II: Treatment Experienced, 1 to 2 Years of Age; Week 12 time point; Test type: Other; % = 50, 95% CI 2-sided [6.8 to 93.2] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort II Week 12, percentage of participants with a >5% decline in absolute CD4 %
Statistical Analysis 3: Comparison: Cohort I: Treatment Experienced, 2 to 6 Years of Age; Week 24 time point; Test type: Other; % = 9.1, 95% CI 2-sided [0.2 to 41.3] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort I Week 24, percentage of participants with a >5% decline in absolute CD4 %
Statistical Analysis 4: Comparison: Cohort II: Treatment Experienced, 1 to 2 Years of Age; Week 24 time point; Test type: Other; % = 25, 95% CI 2-sided [0.6 to 80.6] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort II Week 24, percentage of participants with a >5% decline in absolute CD4 %
Statistical Analysis 5: Comparison: Cohort I: Treatment Experienced, 2 to 6 Years of Age; Week 48 time point; Test type: Other; % = 18.2, 95% CI 2-sided [2.3 to 51.8] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort I Week 48, percentage of participants with a >5% decline in absolute CD4 %
Statistical Analysis 6: Comparison: Cohort II: Treatment Experienced, 1 to 2 Years of Age; Week 48 time point; Test type: Other; % = 50, 95% CI 2-sided [6.8 to 93.2] — Exact Binomial (Clopper-Pearson) confidence intervals for Cohort II Week 48, percentage of participants with a >5% decline in absolute CD4 %

ADVERSE EVENTS:
Time Frame: From entry through off study, at an average of 72 weeks.
Description: At entry, all diagnoses, signs/symptoms and laboratory events were collected. Post-entry, all new diagnoses, signs/symptoms and laboratory events of ≥Grade 1 and all signs/symptoms and laboratory events that led to a change in treatment, regardless of grade, were collected. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used. All eligible participants who initiated study treatment are included.
Arm/Group | Cohort I: Treatment Experienced, 2 to 6 Years of Age | Cohort II: Treatment Experienced, 1 to 2 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/20 | 3/6
Other Adverse Events (participants affected / at risk) | 20/20 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: Treatment Experienced, 2 to 6 Years of Age (N=20) | Cohort II: Treatment Experienced, 1 to 2 Years of Age (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lipase increased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: Treatment Experienced, 2 to 6 Years of Age (N=20) | Cohort II: Treatment Experienced, 1 to 2 Years of Age (N=6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 7 | 3
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Keratosis follicular (Congenital, familial and genetic disorders) | 1 | 0
Ear canal erythema (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 1
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 4 | 3
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0
Eye discharge (Eye disorders) | 2 | 0
Eye pruritus (Eye disorders) | 1 | 0
Eyelid disorder (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 2 | 1
Oral mucosal eruption (Gastrointestinal disorders) | 1 | 0
Palatal disorder (Gastrointestinal disorders) | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Mucosal discolouration (General disorders) | 0 | 1
Pyrexia (General disorders) | 11 | 3
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 1
Acarodermatitis (Infections and infestations) | 2 | 0
Acute sinusitis (Infections and infestations) | 3 | 0
Adenoiditis (Infections and infestations) | 0 | 1
Body tinea (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0
Enterobiasis (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Helminthic infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 5 | 2
Latent tuberculosis (Infections and infestations) | 1 | 0
Lice infestation (Infections and infestations) | 3 | 0
Molluscum contagiosum (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 3 | 3
Otitis media chronic (Infections and infestations) | 1 | 0
Parasitic gastroenteritis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 1
Parvovirus B19 infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 7 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 0
Purulent discharge (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 2 | 0
Sinusitis bacterial (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Tinea capitis (Infections and infestations) | 7 | 0
Tinea faciei (Infections and infestations) | 2 | 0
Tinea manuum (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 2
Toxocariasis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Varicella (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Mucosal excoriation (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 3
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 7 | 1
Blood bicarbonate decreased (Investigations) | 18 | 5
Blood bilirubin increased (Investigations) | 3 | 0
Blood calcium increased (Investigations) | 1 | 1
Blood cholesterol increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose decreased (Investigations) | 7 | 1
Blood glucose increased (Investigations) | 12 | 3
Blood pH decreased (Investigations) | 1 | 0
Blood pH increased (Investigations) | 1 | 1
Blood phosphorus decreased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 2 | 0
Blood potassium increased (Investigations) | 2 | 3
Blood pressure diastolic increased (Investigations) | 4 | 3
Blood pressure systolic increased (Investigations) | 2 | 3
Blood sodium decreased (Investigations) | 14 | 4
Blood sodium increased (Investigations) | 1 | 1
Breath sounds abnormal (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 6 | 5
International normalised ratio increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 4 | 1
Low density lipoprotein increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 9 | 3
Platelet count decreased (Investigations) | 1 | 2
Prothrombin time prolonged (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 2
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Failure to thrive (Metabolism and nutrition disorders) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Hypotonia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 3 | 0
Motor developmental delay (Nervous system disorders) | 0 | 1
Speech disorder developmental (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Penile rash (Reproductive system and breast disorders) | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 6
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 2 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the slow rate of accrual and the challenging accrual into the youngest cohort, enrollment was stopped early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01504841/Prot_001.pdf
  • Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT01504841/SAP_000.pdf